CLINICAL TRIAL: NCT02536482
Title: Tolerability to a New Free Amino Acid-based Formula in Children With Cow's Milk Protein Allergy
Brief Title: Free Amino Acid-based Formula to Treat Children Cow's Milk Protein Allergy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Edetec Indústria Alimentícia S.A. (Industry)
Collaborators: Faculdade de Ciências Médicas de Minas Gerais (Other); Federal University of Minas Gerais (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U1111-1173-4156
Record Dates: First submitted 2015-08-20; First posted 2015-08-31 (Estimated); Last update posted 2015-08-31 (Estimated); Status verified 2015-08

CONDITIONS: Cow's Milk Allergy
MeSH Terms: conditions — Milk Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Amix (Experimental): Dietary supplement. The formula is based in free amino-acid to treat children with cow's milk allergy. The children should have a minimum consumption of 400 mL, daily.
  Interventions: Dietary Supplement: Amix

INTERVENTIONS:
Dietary Supplement: Amix — Treat the children with cow's milk allergy for 5 months.

SUMMARY:
It is a study to assess the tolerance to a new commercially available infant formula in children affected by Cow's Milk Allergy.

DETAILED DESCRIPTION:
In the present study, the children will be followed-up during the treatment with the new formula for Cow's Milk Allergy. They will have monthly doctor's appointment, when the weight, height and symptoms will be evaluated, by a questionnaire and a physical examination.

ELIGIBILITY:
Inclusion Criteria:

* Children with cow's milk allergy

Exclusion Criteria:

* Children without cow's milk allergy

Ages: 1 Day to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2013-08; Primary Completion 2015-02 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Study to assess the allergic symptoms, using a questionnaire. | 5 months
  The allergic symptoms were assessed every month, by using a questionnaire. The parents, during the medical appointment, answered "yes" or "no" according to the presented symptoms: cutaneous (atopic dermatitis and urticaria), gastrointestinal (vomiting, diarrhea constipation and bloody stools ) and respiratory. At the end of the study the children were evaluated if they tolerated the formula, it was observed by the symptoms remission.

SECONDARY OUTCOMES:
Weight assessment, using a digital infant scale | 5 months
  Every medical appointment the doctor measured the weight, by using a digital infant scale. The values were plotted in the software WHO Anthro. A curve weight/age was obtained and the children's weight were compared to the standard population's weight, by the z-score.
Height assessment, using an infantometer | 5 months
  Every medical appointment the doctor measured the height by using a digital infant scale. The values were plotted in the software Anthro. A curve height/age was obtained and the children's height were compared to the standard population's height, by the z-score.
Head circumference, using an infant tape measure | 5 months
  Every medical appointment the doctor measured the head circumference by using a infant tape measure. The values were plotted in the software Anthro. A curve head circumference/age was obtained and the children's head circumference were compared to the standard population's head circumference, by the z-score.

CONTACTS AND LOCATIONS:
Overall Officials: Wendel O Afonso, Master, Study Director — UFMG

REFERENCES:
- [Derived] Amari S, Shahrook S, Namba F, Ota E, Mori R. Branched-chain amino acid supplementation for improving growth and development in term and preterm neonates. Cochrane Database Syst Rev. 2020 Oct 2;10(10):CD012273. doi: 10.1002/14651858.CD012273.pub2. PMID 33006765